CLINICAL TRIAL: NCT04141683
Title: Prognostic Implication of Right Ventricular Contractile Reserve in Patients With Functional Tricuspid Regurgitation
Brief Title: Right VEntricular Contractile ReSERVE in Functional Tricuspid Regurgitation
Acronym: RESERVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Other Study IDs: RESERVE
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: tricuspid regurgitation; heart failure; right heart; stress echocardiography; tricuspid repair; tricuspid replacement
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure | interventions — Echocardiography, Stress; Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stress Echocardiography — Dynamic stress echocardiography using a cycle ergometer on a semi supine exercise table.
Diagnostic Test: Pressure volume loop analysis — Pressure volume loop analysis unsing conductance catheter measurements during right heart catheterization.
Procedure: Tricuspid valve repair or replacement — Tricuspid valve repair or replacement using a surgical or interventionale approach according to local heart team recommendation and patients' preference.

SUMMARY:
Aim of the study is to investigate the prognostic value of right ventricular contractile reserve in patients with functional tricuspid regurgitation undergoing tricuspid valve repair or replacement.

DETAILED DESCRIPTION:
Chronic volume overload in patients with severe tricuspid regurgitation (TR) leads to right ventricular (RV) dilatation, fibrosis and eventually failure. RV dysfunction is an important determinant of mortality in patients undergoing tricuspid valve surgery.

Aim of the current study is to investigate the prognostic utility of right ventricular contractile reserve in patients with severe TR undergoing surgical or interventional tricuspid valve repair or tricuspid valve replacement.

RV contractile reserve will be assessed using semi-supine bicycle stress echocardiography.

Echocardiographic parameters are prone to altered loading conditions, such as volume overload. Load independent RV contractility can only be measured using invasive pressure-volume-loop (PVL) analysis. Therefore RV PVL analysis will be done using conductance catheter in a subset of patients who undergo right heart catheterization for clinical evaluation of pulmonary hypertension. Aim of this sub study is the validation of non-invasively derived RV contractile reserve with load independent markers of intrinsic RV contractility.

ELIGIBILITY:
Inclusion Criteria:

* Severe functional tricuspid regurgitation.
* Planned surgical or interventional tricuspid valve repair or replacement.
* Able to cycle on a semisupine tilting exercise table.
* Informed consent.

Exclusion Criteria:

* Coronary artery disease with significant ischemia.
* Unstable Angina.
* Myocardial infarction <4 month prior to inclusion.
* Concomitant valvular heart disease (aortic, mitral or pulmonary valve) > mild-moderate.
* Constrictive pericarditis.
* Malignant disease with a life expectancy < 12 months.
* Pregnancy.
* Insufficient image quality on echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with severe functional tricuspid regurgitation planned for surgical or interventional tricuspid valve repair or replacement.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Death or heart failure hospitalization | 6-12 month
  Death or heart failure hospitalization according to right ventricular contractile reserve.

SECONDARY OUTCOMES:
Death | 6-12 month
  Death according to right ventricular contractile reserve.
Cardiovascular Death | 6-12 month
  Cardiovascular Death according to right ventricular contractile reserve.
Heart Failure Hospitalization | 6-12 month
  Heart Failure Hospitalization according to right ventricular contractile reserve.
Intrinsic RV contractility | Baseline
  Correlation of RV contractile reserve with the slope of invasively derived right ventricular end systolic elastance.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lurz, MD, PhD, Principal Investigator — University of Leipzig
Locations (1):
- Heart Center Leipzig at Leipzig University, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No